CLINICAL TRIAL: NCT06438679
Title: A Single-centric Prospective Single-arm Study of 3T Therapy in the Treatment of MDA5-positive Dermatomyositis
Brief Title: 3T Therapy in the Treatment of MDA5-positive Dermatomyositis
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB2024-0285
Record Dates: First submitted 2024-05-13; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-02

CONDITIONS: Dermatomyositis
Keywords: MDA5; dermatomyositis; 3T therapy; effectiveness
MeSH Terms: conditions — Dermatomyositis | interventions — tofacitinib; Tacrolimus; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 3T therapy arm (Experimental): This is a single arm experiment
  Interventions: Drug: Tofacitinib 5 MG

INTERVENTIONS:
Drug: Tofacitinib 5 MG — Tofacitinib 5mg BID+thalidomide 50mg BID+tacrolimus 0.1mg/kg QD per oral
  Other Names: tacrolimus; thalidomide

SUMMARY:
The goal of this clinical trial is to learn if a combination of tacrolimus, tafocitinib and thalidomide (3T therapy) works to treat severe MDA5 positive dermatomyositis in adults. It will also learn about the safety of 3T therapy. The main questions it aims to answer are:

Does 3T therapy prolong the overall survival time of MDA5 positive dermatomyositis? What medical problems do participants have when taking 3T therapy?

Participants will:

Take 3T therapy every day for 12 months Visit the clinic once every 2 weeks for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above at the time of screening
* Diagnosis of MDA5-positive dermatomyositis (EULAR/ACR) during screening, and the following 3 items are met at the same time:

  1. The MDA5 titer during screening is ++ or +++;
  2. Mild or above decrease in pulmonary diffusing function at screening and baseline;
  3. Interstitial extravasation seen on chest CT at screening and baseline
* Agree to receive highly effective contraception or sterilized
* Subjects are willing and able to comply with study visits and related procedures
* Subjects have the ability to understand the research requirements and procedures, voluntarily participate in clinical trials and sign the ICF

Exclusion Criteria:

* Have received any drug in 3T treatment in the past, but had poor response (including treatment failure or unacceptable treatment-related adverse reactions)
* Have received lenalidomide, cyclosporine, or other highly selective or pan-selective JAK inhibitors such as lenalidomide or cyclosporine or other highly selective or pan-selective JAK inhibitors such as baricitinib within 2 weeks before visit D1 or within 5 drug half-lives (if known) agent.
* Have received treatment with an immune cell depleting agent (such as rituximab) within 6 months before the D1 visit.
* Have received any investigational drug/treatment within 4 weeks or 5 drug half-lives (if known) before visit D1, whichever is longer.
* Known or suspected history of immunosuppression/deficiency (including but not limited to invasive opportunistic infections such as aspergillosis, coccidioidomycosis, histoplasmosis, AIDS, listeriosis, even if the infection has resolved) within 6 months prior to visit D1, or there are unusually frequent recurring or persistent infections.
* There is a history of malignant tumors within 5 years before the D1 visit (except for completely cured cervical carcinoma in situ or non-metastatic cutaneous squamous cell carcinoma or basal cell carcinoma or thyroid malignant tumors or other malignant tumors considered by the researcher to be amenable to 3T treatment).
* Positive hepatitis B surface antigen (HBsAg) during screening; or positive hepatitis B core antibody (HBcAb) and positive HBV-DNA; or positive hepatitis C antibody and positive HCV ribonucleic acid (RNA) polymerase chain reaction; or human immune HIV-deficiency virus (HIV) serology was positive.
* Subjects with active tuberculosis, latent tuberculosis, or a history of non-tuberculous mycobacterial infection at the time of screening.
* Have a history of systemic hypersensitivity reaction to any drug or matrix or excipient in 3T therapy.
* Have been vaccinated within 12 weeks before the D1 visit, or plan to receive a live (attenuated) vaccine during the study.
* Pregnant or lactating women, or subjects who plan to become pregnant or lactating during the study.
* Any other circumstances in which the researcher determines that it is not appropriate to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | 26 weeks
  The overall survival rate at the end of observation
Overall TE incidence | 26 weeks
  The overall treatment associated adverse effects incidence during the clinical trial

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang University School of Medicine Second Affiliated Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided